CLINICAL TRIAL: NCT04253405
Title: Multicentric Randomized Controlled Pilot Study Comparing High Flow Nasal Cannula Versus NonInvasive Positive Pressure Ventilation in Acute Respiratory Failure in Patients With Pulmonary Fibrosis (RENOVATE Fibrosis)
Brief Title: RENOVATE Fibrosis:HFNC Versus NIPPV in Acute Respiratory Failure in Patients With Pulmonary Fibrosis
Acronym: Fibrosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study impacted by the COVID-19 pandemic:
  * slow recruitment rate
  * budget constrains
Sponsor: Hospital do Coracao (Other)
Collaborators: Ministry of Health, Brazil (Other Government); Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IP-HCOR/RENOVATEfibrose
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Acute Respiratory Failure; Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis | interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: 1:1 randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Flow Nasal Cannula (HFNC) (Active Comparator): The HFNC (Airvo2 Fisher & Paykel, Auckland, New Zealand) consists of an apparatus that allows adjustable FiO2 from 21 to 100% and delivers flow up to 60 L/ min.
  Interventions: Device: High Flow Nasal Catheter
- Non-invasive positive pressure ventilation (NIPPV) (Active Comparator): NIPPV will be performed using the devices available on centers. Both a dedicated NIPPV device or an invasive mechanical ventilator with NIPPV mode are accepted. The interface should be an oronasal or full face mask.
  Interventions: Device: Noninvasive positive pressure ventilation (NIPPV)

INTERVENTIONS:
Device: High Flow Nasal Catheter — HFNC will be delivered through AIRVO2. FiO2 from 21 to 100% and heated humidified gas flow up to 60 l / min with temperature of the circuit maintained at 37 degrees.
  Oxygen flow will be offered through a humidified nasal catheter. Flow and FiO2 will be titrated according to the protocol to maximize the patient´s comfort and SpO2
  Other Names: Optiflow; Airvo; trans-nasal insufflation; Nasal High Flow; High Flow Nasal Cannula
  Arms: High Flow Nasal Cannula (HFNC)
Device: Noninvasive positive pressure ventilation (NIPPV) — NIPPV will be performed using a facial mask (either oronasal or full face). NIPPV will deliver pressures and FiO2 according to the protocol.
  Other Names: BiPAP; Non-invasive ventilation; Non-invasive positive pressure ventilation
  Arms: Non-invasive positive pressure ventilation (NIPPV)

SUMMARY:
A pilot multicentric randomized controlled study investigating the feasibility of recruiting 50 pulmonary fibrosis patients in acute respiratory failure within18 months. Additionally, exploratory efficacy and safety outcomes will be evaluated.

DETAILED DESCRIPTION:
RENOVATE Fibrosis will recruit patients with pulmonary fibrosis in acute respiratory failure to be randomized to HFNC or NIPPV. Efficacy and safety outcomes measured are dyspnea variation, physiological variables (pCO2, respiratory rate, oxygenation), comfort, endotraqueal intubation rate, mortality in 28 and 90 days.

ELIGIBILITY:
Inclusion Criteria: Sequential adult patients 18 years of age or older admitted to the hospital with pulmonary fibrosis and acute onset of respiratory failure that meets criteria A and B bellow.

A. Pulmonary fibrosis will be defined by all of the criteria below:

* presence of Velcro-type crackles on physical examination
* imaging compatible with pulmonary fibrosis
* diffuse disease on imaging

B. Acute respiratory failure (ARF) will be defined by hypoxemia evidenced by SpO2 <90% or PaO2 <60 mmHg in room air and at least two of the criteria below within the last four weeks:

* worsening dyspnea
* worsening breathing effort
* worsening gas exchange (worsening SpO2 or paO2)
* worsening respiratory rate, above 25 irpm

Exclusion Criteria:

* Pulmonary fibrosis secondary to progressive massive fibrosis (silicosis), or any other tumor form of fibrosis;
* Significant pulmonary arterial hypertension characterized by: Right ventricular failure on Doppler echocardiogram or Cardiac index <2L / min / m2 in catheterization of right chambers;
* Pneumothorax or extensive pleural effusion as the main determinant of ARF in the assessment of the attending physician;
* Cardiogenic pulmonary congestion as the main determinant of IRPA in the assessment of the attending physician;
* Presence of delirium or non-cooperation at the time of randomization;
* Anatomical facial abnormalities;
* Incoercible vomiting or hypersecretion of the airways;
* Use of continuous VNIPP or HFNC for more than 8h before randomization;
* pregnancy;
* Refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2021-08-09 (Actual)

PRIMARY OUTCOMES:
Recruitment feasibility | 18 months
  Recruitment of 50 pulmonary fibrosis patients in acute respiratory failure in 18 months

SECONDARY OUTCOMES:
Dyspneia variation (Borg scale) | 7 days
  Borg scale
Respiratory frequency variation | 7 days
  Respiratory rate
oxygen saturation/fraction of inspired oxygen (SpO2/FiO2) variation | 7 days
  Oxygen index
Carbon dioxide arterial partial pressure (PaCO2) variation | 7 days
  CO2 variation

OTHER OUTCOMES:
Comfort visual analog scale variation | 7 days
  Confort scale
Endotracheal intubation (ETI) rate | 7 days
  Endotracheal intubation
Mortality | 28 days
  Mortality in 28 days
Mortality | 90 days
  Mortality in 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Leticia Kawano-Dourado, MD, Principal Investigator — Hospital do Coração; Israel Maia, MD, Principal Investigator — Hospital do Coração
Locations (6):
- Brazil (6):
  - Hospital UNIMED Vitória, Vitória, Espírito Santo
  - Hospital de Brasilia (HOBRA), Brasília, Federal District
  - Hospital Nereu Ramos, Florianópolis, Santa Catarina
  - Instituto de Cardiologia Dante Pazanese, São Paulo, São Paulo
  - Hospital do Coracao, São Paulo
  - InCor - Hospital das Clinicas da Faculdade de Medicina da USP, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Data sharing plan - under construction
Supporting Information: Study Protocol, SAP, ICF
Time Frame: In 8 months
Access Criteria: Publication